CLINICAL TRIAL: NCT06967844
Title: Effects of Simultaneous Versus Sequential Motor-cognitive Task Training on Balance and Coordination Among Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/60
Record Dates: First submitted 2024-12-12; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Balance; Cognitive Functions
Keywords: balance; coordination; dual-task performance; Simultaneous Motor-cognitive task training; Sequential Motor-cognitive task training; cognition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simultaneous motor-cognitive task training (Experimental): It includes elderly individuals receiving simultaneous motor-cognitive task training for balance, coordination, dual-task performance and cognition for 40 min duration (6 weeks with 2 sessions per week).
  1. Walking while counting walk 5 meters while counting backward by ones walk 10 meters while counting backward by threes walk 15 meters while counting backward by sevens
  2. Balancing on one foot while naming and solving puzzle stand on one foot for 20 seconds while naming animals stand on one foot for 30 seconds while solving simple puzzle stand on one foot for40 seconds while solving complex puzzle
  3. Ball toss and recall toss a ball at 3 meters while recalling three word list toss a ball at 5 meters while recalling five word list toss a ball at 7 meters while recalling seven word list
  Interventions: Procedure: Simultaneous motor-cognitive task training
- Sequential motor-cognitive task training (Active Comparator): It includes elderly individuals receiving sequential motor-cognitive task training for balance, coordination, dual-task performance and cognition for 20 minutes duration each (motor and cognition training) with a 20 min rest in between (6 weeks with 2 sessions per week).
  Motor-training :
  1. Balancing on one foot standing on one foot for 10 seconds standing on one foot for 20 seconds standing on one foot for 30 seconds
  2. Heel-to-toe walk walk heel to toe 5 meters walk heel to toe 10 meters walk heel to toe 15 meters
  3. Leg swings 10 swings per leg 15 swings per leg 20 swings per leg
  Cognitive-training :
  1. Memory games recall three word list recall five word list recall seven word list
  2. Problem-solving tasks simple arithmetic problems moderate level arithmetic problems difficult arithmatic problems
  Interventions: Procedure: Sequential motor-cognitive task training

INTERVENTIONS:
Procedure: Simultaneous motor-cognitive task training — 16 sessions (2 sessions per week) for 8 weeks, 40 min per session
  1. walking while counting walk 5, 10 and 15 meters while counting backward by ones, threes and sevens
  2. balancing on one foot while naming or solving puzzles stand on one foot for 10, 20 and 30 seconds while naming animals. solving simple and complex puzzles
  3. ball toss and recall toss ball at 3, 5 and 7 meters distance while recalling three-word, five-word and seven-word lists
  Arms: Simultaneous motor-cognitive task training
Procedure: Sequential motor-cognitive task training — 16 sessions (2 sessions per week), for 8 weeks, 20+20 min per session with 20 min break in between
  motor training
  1. Standing on one foot standing on one foot for 10, 20 and 30 seconds
  2. Heel to toe walk walking heel to toe for 5, 10 and 15 meters
  3. Leg swings 10 swings, 15 swings and 20 swings per leg cognitive training
  4. Memory games recall three-word, five-word and seven-word lists
  5. Problem solving tasks simple, moderate and difficult arithmetic problems
  Arms: Sequential motor-cognitive task training

SUMMARY:
A randomized control trial will be done on elderly individuals in Community Homes of Rawalpindi/Islamabad. Motor-cognitive impairments impact the life of elderly individuals. The purpose of the study is to determine the effects of simultaneous versus sequential motor-cognitive task training on balance, coordination, dual task performance and cognitive functions using the Berg Balance Scale, Mini Mental State Examination, Fall Efficacy Scale and time up and go test, The Simultaneous Motor-cognitive task traning includes activities like walking while counting, balancing on one foot while naming or solving puzzles, and ball toss with recall for forty minutes. The sequential motor-cognitive task training includes standing on one foot, heel-to-toe walk, and leg swings for 20 minutes; and after 20 min rest time followed by memory games and problem-solving tasks for 20 minutes. 12 sessions for 6 weeks will be given.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* MMSE scoring 24 or higher
* BBS scoring 41-56

Exclusion Criteria:

* cardio, neurological, musculoskeletal, and psychiatric problems.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Balance | 6 weeks
  Berg Balance Scale will be used to assess balance. It has total number of 14 items, and total score of 56
Dual task performance | 6 weeks
  dual task performance will be assessed using Timed up and go test.
Cognition | 6 weeks
  mini-mental state examination (total number of items is 11, total score is 30)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan